CLINICAL TRIAL: NCT01127100
Title: Gabapentin Versus Transdermal Fentanyl Matrix (TDF) for Chronic Neuropathic Pain (of Radicular Origin): A Multicenter Randomized, Parallel Group, Rater Blinded, Non-inferiority Trial
Brief Title: Gabapentin Versus Transdermal Fentanyl Matrix for Chronic Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Asan Medical Center (Other); Inje University (Other); Chonnam National University Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Dankook University (Other)
Responsible Party: Principal Investigator, Jae Hyup Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neuropathic pain 2010
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Neuropathic Pain; Spinal Stenosis
Keywords: neuropathic pain; gabapentin; transdermal fentanyl matrix; multicenter; non-inferiority trial
MeSH Terms: conditions — Neuralgia; Spinal Stenosis | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transdermal fentany matrix (Experimental): Transdermal fentanyl matrix is second-line medication on the neuropathic pain but gabapentin is the first-line medication. So, transdermal fentanyl matrix is experimental arm and gabapentin is active comparator arm.
  Interventions: Drug: transdermal fentanyl matrix, gabapentin
- gabapentin (Active Comparator): Gabapentin is the first-line medication in neuropathic pain. So, gabapentin is active comparator in this study and transdermal fentanyl matrix is experimental.
  Interventions: Drug: transdermal fentanyl matrix, gabapentin

INTERVENTIONS:
Drug: transdermal fentanyl matrix, gabapentin — transdermal fentanyl matrix: during 1st to 6th days, 12ug/h of fentanyl matrix will be applied. During 7th to 28th days, the dosage of fentanyl matrix will be increased until the pain score decrease not more than 2 every 6 days. The maximal dosage is 100ug/h. During 29th to 56th days, the dosage will be maintained.
  Gabapentin: the 1st day, 300mg hs, the 2nd day, 300mg bid, the 3th to 4th days, 300mg tid, the 5th to 6th days, 300mg-300mg-600mg the 7th to 28 days, the dosage will be increased until the pain score decreased not more than 2 and the maximal dose is 2400mg per day. During 29th to 56th days, the dosage will be maintained.

SUMMARY:
Gabapentin is a first line medication and fentanyl is second line medication in neuropathic pain. But, there is no head to head study on the efficacy of those medication in neuropathic pain.

The hypothesis of this study is that the efficacy of the transdermal fentanyl matrix is not inferior to the gabapentin in neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* patients are 20 years of age or older
* patients had chronic pain for more than 3 months and average pain score for last 3 days is not less than 4 (NRS)
* neuropathic pain caused by the spinal stenosis (radiating pain, motor or sensory change
* positive MRI finding or radiculopathy was confirmed by the EMG/NCS or not less than 12 points in the S-LANSS score assessment
* patients who can make out the questionnaire
* patients have agreed with the informed consent

Exclusion Criteria:

* patients who have experience with gabapentin, pregabalin, fentanyl matrix, long-acting strong opioid (CR oxycodone, SR morphine)
* patients who have other causes of neuropathy such as hypothyroidism, Vit B12 deficiency, connective tissue disease, etc.
* patients who have other disease which causes more pain compared with neuropathic pain
* patients with a history of drug or alcohol abuse
* patients who are pregnant or have the possibility of pregnancy
* patients who are unable to use a transdermal system due to skin disease
* patients with a serious mental disease
* patients with a history of hypersensitivity to opioid analgesics
* patients with a chronic pulmonary disease or respiratory depression
* patients combined with industrial accidents or traffic accidents
* at investigator's discretion, any condition where a subject cannot take part in the clinical study on the ground of warning, cautions, and prohibition in study investigator's brochure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity difference between gabapentin used group and transdermal fentanyl matrix used group | Visit1 (Day 1), Visit 2 (Day 22-36), Vist3 (Day 50-64)
  Post-treatment pain intensity scores will be used to determine the percentage of pain intensity difference between gabapentin used group and transdermal fentanyl matrix used group.

SECONDARY OUTCOMES:
Differences of Oswestry Disability Index score, SF-36, BDI score, investigator and patients global assessment between gabapentin used group and transdermal fentanyl matrix used group | Visit 1(Day 1), Visit 2(Day 22-36), Visit 3 (Day 50-64)
  Post-treatment secondary efficacy assessments will be used to determine the percentage of difference and secondary efficacy assessments included the following. 1. Korean Oswestry Disability Index score, Korean-Short-Form 36, Beck Depression Index score, investigator and patients global assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hyup Lee, MD, PhD, Principal Investigator — Seoul National University, College of Medicine, Department of Orthopedic Surgery, SMG-SNU Boramae Medical Center
Locations (1):
- Seoul National University, College of Medicine, Department of Orthopedic Surgery, SMG-SNU Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hwang CJ, Lee JH, Kim JH, Min SH, Park KW, Seo HY, Song KS. Gabapentin versus Transdermal Fentanyl Matrix for the Alleviation of Chronic Neuropathic Pain of Radicular Origin: A Randomized Blind Multicentered Parallel-Group Noninferiority Trial. Pain Res Manag. 2019 Feb 4;2019:4905013. doi: 10.1155/2019/4905013. eCollection 2019. PMID 30863474